CLINICAL TRIAL: NCT06941974
Title: Partnering With Antenatal Navigators to Transform Health in Pregnancy
Acronym: PATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Lynn M Yee, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00218597; R01MD020130 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-04-24 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Maternal Morbidity; Antenatal Health; Neonatal Morbidity; Retention in Care; Prenatal Care
MeSH Terms: interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: There will be two cohorts: One cohort will be provided intensive, individualized, one-on-one navigation services from early pregnancy (before 20 weeks of gestation) through 2 weeks postpartum. The second cohort will receive usual care. Both cohorts will be followed through 9 months postpartum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigation Group (Experimental): Pregnant participants who are randomized to receive PATH patient navigation will be assigned to a patient navigator. The patient navigator will meet with the patient in early pregnancy for introductions, education, and assessing factors that influence health and access to care. The patient navigator will offer support and resources (e.g., appointment coordination and scheduling, communication with clinical team, transportation, community referrals, support for mental health, support for other non-medical needs, etc.). The navigator will provide support and continue linkage to resources through 2 weeks postpartum.
  Interventions: Behavioral: Patient Navigation Program
- Non-navigation Group (No Intervention): No navigation will be provided; pregnant participants will receive usual care.

INTERVENTIONS:
Behavioral: Patient Navigation Program — PATH navigation is an antenatal patient navigator program designed to reduce barriers to care, enhance access, improve self-efficacy and knowledge, and improve multiple perinatal health outcomes. PATH navigation is a flexible, multi-pronged, patient-centered program with the capacity to evolve with patient needs and preferences. Early in pregnancy, navigators will establish themselves as a non-medical resource and will introduce PATH as a program designed to help inform, support, and connect patients during pregnancy. Navigators will review screen and address supportive and adverse non-medical needs, facilitate communication, perform logistical support, provide advocacy and bridge communication with clinical teams, and perform health education. Navigation services will be tailored to individual medical, psychosocial, or logistical complexity.
  Arms: Navigation Group

SUMMARY:
The Partnering with Antenatal Navigators to Transform Health in Pregnancy (PATH) study aims to evaluate whether an antenatal patient navigation program improves maternal health, neonatal health, pregnant women's experiences, and health care utilization outcomes among low-income pregnant women and their neonates. Patient navigation is an individualized, barrier-focused, longitudinal, patient-centered intervention that offers support for a defined set of health services. In this randomized controlled trial, pregnant women who are randomized to receive antenatal patient navigation will be compared to pregnant women who are randomized to receive usual care. Navigators will support pregnant women from before 20 weeks of gestation through 2 weeks postpartum. The PATH intervention will be grounded in understanding and addressing factors that influence health and access to care in order to promote self-efficacy, enhance access, and sustain long-term engagement.

The main objectives of the study are to:

1. Evaluate whether PATH, compared to usual care, improves maternal health outcomes. We hypothesize the PATH model of antenatal patient navigation for low-income women will reduce the incidence of a composite of adverse maternal outcomes, all of which are known to be increased among women with barriers to care.
2. Evaluate whether PATH, compared to usual care, improves perinatal health outcomes. We hypothesize PATH will reduce the incidence of a composite of adverse perinatal outcomes. We will also investigate neonatal/pediatric health care utilization.
3. Evaluate patient, clinician, navigator, and healthcare system experiences with PATH in preparation for widespread implementation and dissemination of the PATH obstetric navigation model. This aim will be accomplished through investigating patient-reported outcomes, completing qualitative and process mapping interviews with navigated participants, and completing qualitative and process mapping interviews with clinicians, navigators, and health administrators.

DETAILED DESCRIPTION:
In the US, high rates of maternal morbidity are urgent public health concerns. Limited access to health care combined with other non-medical challenges generate greater risk of adverse maternal and neonatal outcomes for women with low income. High-quality antenatal care supports optimal health, yet typically fails to meet the needs of some populations, including those with lower incomes. Improving the health of pregnant women in a patient-centered manner requires innovative models of care delivery across the spectrum of maternal care. One strategy is patient navigation, a longitudinal, barrier- focused, patient-centered intervention that offers support for health services. Our prior work has included the study of patient navigation for low-income postpartum women, finding that assignment to a navigator improves the receipt of postpartum care and the successful transition to primary care. Although antenatal care is an ideal setting for patient navigation, the benefits of antenatal patient navigation for overall maternal and perinatal health have not been rigorously evaluated in randomized trials. There has been no study of antenatal patient navigation as a comprehensive, wraparound service to improve a wide range of pregnancy outcomes.

This randomized controlled trial aims to test the efficacy of an innovative antenatal care patient navigation model that extends and expands care for low-income pregnant women via the Partnering with Antenatal Navigators to Transform Health in Pregnancy (PATH) Trial. We will randomize nulliparous pregnant women with low income to receive antenatal patient navigation via the PATH program versus usual antenatal care. Participants randomized to receive PATH navigation will receive intensive, individualized patient navigation services throughout pregnancy. As a multilevel, multidomain, intervention, PATH navigation is grounded in understanding and addressing approaches to promote self-efficacy, enhance access, support communication, and sustain healthcare engagement. The PATH navigation program is a comprehensive antenatal patient navigator program which is guided by principles of barrier ascertainment and reduction, promotion of self-efficacy and health literacy skills, facilitation of communication, and enhancing antenatal care access. PATH navigators will incorporate best practices regarding non-medical needs assessment, motivational interviewing, health education, and capacity-building health behavior support.

The study will enroll and randomize 550 to 600 pregnant women, ages 16 and over, who have not had a previous live birth and who have publicly funded prenatal care or have low income. Participants assigned to navigation will be provided intensive, individualized, one-on-one navigation services from enrollment (at less than 20 weeks of gestation) through 2 weeks postpartum. All participants will undergo surveys, interviews, and medical record reviews at 5 study visits from enrollment (<20 weeks of gestation) through 9 months postpartum. Visits will occur at the following intervals: before 20 weeks (V1), 28-32 weeks of gestation (V2), at the time of hospitalization for delivery (V3), 6-12 weeks postpartum (V4), and 9 months postpartum (V5).

Aim 1 will evaluate whether PATH, compared to usual care, improves a composite of maternal adverse outcomes (including hypertensive disorders, preterm birth, postpartum hemorrhage, severe maternal morbidity, maternal mortality). Sub-Aim 1 aims to evaluate whether PATH, compared to usual care, improves effective maternal healthcare utilization (antenatal hospital use, Adequacy of Prenatal Care Utilization index, postpartum care/admission). Aim 2 will evaluate whether PATH, compared to usual care, improves a composite of perinatal adverse outcomes (including neonatal intensive care unit admission, low birthweight, small- and large-for-gestational age, perinatal death). Sub-Aim 2 aims to evaluate whether PATH, compared to usual care, improves effective neonatal/pediatric healthcare utilization (neonatal length-of-stay, neonatal hospital utilization, and pediatric care attendance). Exploratory Aims 1 and 2 will evaluate whether PATH's efficacy varies by different demographic factors (e.g. age), or chronic disease status.

Aim 3 will evaluate patient, clinician, navigator, and health system experiences with PATH in preparation for widespread implementation and dissemination of the PATH obstetric navigation model. This aim is guided by implementation science principles and will be accomplished via serial collection of patient-reported outcomes, individual interviews, and process mapping exercises. Specifically, Aim 3a will compare patient-reported outcomes, including perceived health status, quality of life, patient activation, stress level, and self-efficacy, for women who receive PATH navigation versus usual care. Aim 3b will use qualitative and process mapping methods among approximately 50 participants assigned to PATH to understand participants' engagement, feedback, pregnancy experience, antenatal care processes, and satisfaction with the level of social and medical care received with patient navigation. Aim 3c will similarly use qualitative and process mapping methods with approximately 20 clinicians, navigators, and health system administrators to understand the extent to which PATH facilitated clinical, administrative, and health system needs, as well as lessons for future program implementation, including the relative benefits of discrete elements of the PATH intervention.

The PATH Trial will fill a significant evidence gap by demonstrating whether antenatal patient navigation among low-income pregnant women, who are disproportionately at risk for adverse outcomes, is an effective strategy to improve perinatal health. The expected outcome of this project is to generate the empiric evidence needed to understand the effect of antenatal patient navigation and to plan for an optimized package of successful implementation strategies to prepare for broad dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation <20 weeks of gestation
* Nulliparous: no prior pregnancies ≥20 weeks excluding terminations
* Low income (public insurance or residence in a neighborhood in which >10% of household incomes are <125% of federal poverty line
* Ability to speak and read English or Spanish
* Established patient at one of practices associated with Northwestern Medical Group
* Age 16 years or older

Exclusion:

* Intent to transfer care to an outside institution
* Prior enrollment in PATH
* Concurrent enrollment in a study with competing aims/intervention

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Maternal adverse outcome composite (Aim 1 primary outcome) | Enrollment through delivery hospitalization, an average of 28 weeks
  Frequency of maternal composite, which includes hypertensive disorders of pregnancy, preterm birth, postpartum hemorrhage, severe maternal morbidity, or maternal mortality. Components of the primary outcome will also be examined as a score and individually as secondary outcomes (see below).
Neonatal adverse outcome composite (Aim 2 primary outcome) | At birth/delivery
  Frequency of the neonatal composite, which includes neonatal intensive care unit (NICU) admission, low birthweight, small-for-gestational-age (SGA), large-for-gestational-age (LGA) status, and/or perinatal death. Components of the composite outcome will also be examined as a score and individually as secondary outcomes (see below).

SECONDARY OUTCOMES:
Hypertensive disorder of pregnancy (component of primary outcome) | Enrollment through delivery hospitalization, an average of 28 weeks
  Frequency of de novo hypertensive disorder of pregnancy, including gestational hypertension, preeclampsia with or without severe features, superimposed preeclampsia on chronic hypertension, eclampsia, or HELLP syndrome
Preterm birth (component of primary outcome) | Enrollment through delivery hospitalization, an average of 28 weeks
  Frequency of birth less than 37 weeks of gestation
Postpartum hemorrhage (component of primary outcome) | At birth/delivery
  Frequency of estimated/quantitative blood loss >1000mL (during delivery hospitalization) or blood transfusion
Severe maternal morbidity (component of primary outcome) | Enrollment through delivery hospitalization, an average of 28 weeks
  Frequency of CDC-defined indicators for severe maternal
Maternal mortality (component of primary outcome) | Enrollment through delivery hospitalization, an average of 28 weeks
  Frequency of maternal death (any reason) during pregnancy or the delivery hospitalization
Neonatal intensive care unit admission (component of Aim 2 neonatal composite outcome) | At birth/delivery
  Frequency of admission to the neonatal intensive care unit
Low birthweight (component of Aim 2 neonatal composite outcome) | Immediately post-birth
  Frequency of birth weight <2500g
Small-for-gestational-age (SGA) status (component of Aim 2 neonatal composite outcome) | Immediately post-birth
  Frequency of birth weight <10%ile for gestational age and sex
Large-for-gestational-age (LGA) status (component of Aim 2 neonatal composite outcome) | Immediately post-birth
  Frequency of birth weight >90%ile for gestational age and sex
Perinatal death (component of Aim 2 neonatal composite outcome) | 20 weeks of gestational through birth hospitalization
  Frequency of intrauterine fetal demise (>20 weeks of gestation) or neonatal death (i.e., antenatal, intrapartum, or neonatal death)
Maternal health care utilization: Antenatal hospital utilization | Enrollment through delivery
  Frequency of unanticipated obstetric triage or emergency department visit, or antepartum admission
Maternal health care utilization: Antenatal care adequacy | Enrollment through delivery
  Adequacy of Prenatal Care Utilization Index score
Maternal health care utilization: Postpartum care | Between delivery and 12 weeks after delivery
  Frequency of attendance at a routine postpartum care visit within 12 weeks after delivery
Maternal health care utilization: Postpartum admission or emergency department use | Between delivery and 9 months postpartum
  Frequency of hospital readmission or emergency department use within 9 months of delivery
Neonatal health care utilization: Neonatal length of stay | During birth hospitalization
  Neonatal length of birth hospitalization (days)
Neonatal health care utilization: Neonatal hospital utilization | From birth hospital discharge through 9 months
  Frequency of neonatal emergency department visit or hospital admission
Neonatal health care utilization: Pediatric care attendance | From birth hospital discharge through 9 months
  Frequency of attendance at indicated neonatal/pediatric outpatient care in the recommended time frame in the first 9 months of life
Patient-reported outcome: Global health status | During pregnancy, delivery hospitalization, 6-12 weeks postpartum, and 9 months postpartum
  PROMIS Global Health score
Patient-reported outcome: Health-related quality of life | During pregnancy, delivery hospitalization, 6-12 weeks postpartum, and 9 months postpartum
  Short Form Health Survey score
Patient-reported outcome: Depressive symptoms | During pregnancy, delivery hospitalization, 6-12 weeks postpartum, and 9 months postpartum
  Patient Health Questionnaire-9 score
Patient-reported outcome: Anxiety symptoms | During pregnancy, delivery hospitalization, 6-12 weeks postpartum, and 9 months postpartum
  General Anxiety Disorder-7 score
Patient-reported outcome: Health-related self-efficacy | During pregnancy, delivery hospitalization, 6-12 weeks postpartum, and 9 months postpartum
  PROMIS Self-Efficacy-General score
Patient-reported outcome: Patient activation | During pregnancy, delivery hospitalization, 6-12 weeks postpartum, and 9 months postpartum
  Consumer Health Activation Index score
Patient-reported outcome: Difficulties in pregnancy | During pregnancy, delivery hospitalization, and 6-12 weeks postpartum
  nuMoM2b Difficulties in Pregnancy Scale score
Patient-reported outcome: Pregnancy experiences | 3rd trimester, delivery hospitalization
  nuMoM2b Pregnancy Experience Scale-Brief score
Patient-reported outcome: Stress | During pregnancy, delivery hospitalization, 6-12 weeks postpartum, and 9 months postpartum
  Perceived Stress Scale score
Patient-reported outcome: Satisfaction with care (antenatal and postpartum) | During pregnancy, delivery hospitalization, and 6-12 weeks postpartum
  Prenatal Care Satisfaction Scale score and modified scale for postpartum care satisfaction

OTHER OUTCOMES:
Participant experiences with patient navigation and antenatal care process mapping | Enrollment through delivery hospitalization, an average of 28 weeks
  Participants randomized to receive navigation will complete in-depth qualitative interviews on their experiences with the navigation program. Interviews will address satisfaction with social and medical care received, engagement with the program, antenatal care experience, relationship with the navigator, experience with PATH navigation, and areas for improvement. Interviews will also include process mapping to understand antenatal care processes and PATH's contributions to their optimization
Satisfaction with navigation (interpersonal aspects) | During pregnancy and through 9 months postpartum
  Survey - Patient Satisfaction with Interpersonal Relationship with Navigator Scale (among participants receiving navigation)
Satisfaction with navigation (logistical aspects) | During pregnancy and through 9 months postpartum
  Survey - Patient Satisfaction with Logistical Aspects with Navigator Scale (among participants receiving navigation)
Clinician, navigator, and administrator interviews and process mapping | Through completion of study, an average of 5 years
  Clinicians, navigators, and administrators will complete in-depth interviews and process mapping exercises. Interviews will solicit their input whether PATH is successful, preferred patient navigation elements, and how they perceive PATH to affect patient care. Interviews will also include implementation science-guided process mapping exercises to understand how PATH navigation intersects with system-level healthcare, patient-level needs, and organizational processes.
Navigation intensity and activities | Through completion of study, an average of 5 years
  Mixed methods data on navigation intensity (number of interactions over the duration of intervention performance), types of activities completed for/with participants, types of communication modes used, and types of health care team interactions. Data will be integrated from navigator logs of navigation activities and quarterly in-depth qualitative interviews with the navigators.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn M Yee, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No